CLINICAL TRIAL: NCT03680833
Title: Sentinel Node Detection in Cervical Cancer
Acronym: SLNcxca
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RegionSkaneKKLund2
Record Dates: First submitted 2018-09-14; First posted 2018-09-21 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Sentinel Lymph Node Biopsy

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- prospective cohort study (Other): Prospective cohort study with detection of sentinel lymph nodes followed by a full pelvic lymphadenectomy. Patients will act as their own controls.
  The intervention is the detection and removal of sentinel lymph nodes
  Interventions: Procedure: Sentinel node detection in cervical cancer

INTERVENTIONS:
Procedure: Sentinel node detection in cervical cancer — The study intervention is the injection of tracer followed by detection and removal of sentinel lymph nodes

SUMMARY:
Evaluation of sensitivity of Sentinel lymph nodes for detecting nodal metastases in cervical cancer

DETAILED DESCRIPTION:
Consecutive women with stage 1a2-2a1 cervical cancer scheduled for surgery will be approached for eligibility by defined criteria.

Sentinel nodes will be detected by a combined use of Indocyanine green and Tc99 radiocolloid ( first 75 patients) and for the continuation with either the combined use or the best performing of those tracers.

Technical success rates, adverse events (related study intervention and overall) sensitivity and negative predictive values will be estimated.

An interim analyse will be performed after 34 node positive patients based on the Fleming two stage analyse. The null hypothesis of sensitivity of 85% will be tested against an estimated sensitivity of 95%. At this stage the study may be closed for futility, closed as hull hypothesis is rejected or continued to reach another 28 node positive patients.

As a full pelvic lymphadenectomy will be performed after detection of sentinel nodes patient will act ast their own controls.

ELIGIBILITY:
Inclusion Criteria:

* Women of age 18 years and older at the time of informed consent.
* Women with a pathologically proven cervical carcinoma of any histologic subtype, clinically stage 1a2- 2a1 planned for primary surgery
* Absence of any exclusion criteria

Exclusion Criteria:

* Non consenting patients
* Ongoing pregnancy
* Inability to understand written and/or oral study information
* Who performance status III or more
* Previous lower limb lymphedema
* Surgical contraindication to a laparoscopic approach or lymphadenectomy at surgeons discretion.
* Anesthesiologic contraindication to a laparoscopic approach at the anesthetist's discretion
* Locally advanced disease or intraabdominal/distant metastases at preoperative CT, MRI or ultrasonography
* Radiologically suspect pelvic nodal metastatic disease according to the RECIST criteria (>= 1 node with >=16 mm short axis diameter)
* Allergy to Iodine
* Patients with a known liver disease
* Patients with a significant bleeding disorder or mandatory antithrombotic treatment.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2014-06-15 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sentinel node detection in cervical cancer; Sensitivity and negative predictive values for identifying pelvic nodal disease, See detailed study protocol | 4-5 years
  Detection of Sentinel nodes followed by full pelvic lymphadenectomy

CONTACTS AND LOCATIONS:
Overall Officials: Jan Persson, ass professor, Principal Investigator — Region Skane
Locations (1):
- Department of Gynecology and Obstetrics, Lund, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT03680833/Prot_SAP_000.pdf